CLINICAL TRIAL: NCT05766007
Title: Long-acting Injectable Antipsychotics for Mental Ill-Health in Pregnancy and Postpartum: An Observational Cohort Study
Brief Title: Long-acting Injectable Antipsychotics for Mental Ill-Health in Pregnancy and Postpartum
Acronym: LAMP
Status: Recruiting | Type: Observational
Sponsor: University of Liverpool (Other)
Collaborators: Federal Neuropsychiatric Hospital, Yaba (Unknown); Federal Neuropsychiatric Hospital, Kaduna (Unknown); Neuropsychiatric Hospital, Abeokuta (Unknown); Neuropsychiatric Specialist Hospital, Akure (Unknown); Obafemi Awolowo University Teaching Hospital (Other); Federal Medical Centre, Makurdi (Unknown)
Responsible Party: Sponsor
Other Study IDs: UoL001749
Record Dates: First submitted 2023-01-30; First posted 2023-03-13 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia; Psychosis; Mania; Pregnancy; Drug Exposure in Utero; Drug Exposure Via Breast Milk; Antipsychotic Agents; Breastfeeding
Keywords: mental ill health; pregnancy; postpartum; long-acting injectable antipsychotics; Risperidone; Paliperidone palmitate; Fluphenazine decanoate; Flupentixol decanoate; Zuclopenthixol decanoate
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mania; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dried blood spots and dried breastmilk spots on protein saver cards
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Risperidone: Pregnant or breastfeeding women receiving the long acting injectable form of Risperidone and their babies
- Paliperidone palmitate: Pregnant or breastfeeding women receiving Paliperidone palmitate and their babies
- Flupentixol decanoate: Pregnant or breastfeeding women receiving the Flupentixol decanoate and their babies
- Zuclopenthixol decanoate: Pregnant or breastfeeding women receiving the Zuclopenthixol decanoate and their babies
- Fluphenazine decanoate: Pregnant or breastfeeding women receiving the Fluphenazine decanoate and their babies

SUMMARY:
The goal of this observational study is to learn about how long-acting injectable antipsychotic (LAIA) medications are affected by the changes that take place in the body during pregnancy, and how much an unborn baby is exposed to. The investigators are also interested in the amount of these drugs that enters into breastmilk and taken by babies during breastfeeding.

In addition to their regular clinic visits to receive long-acting mental health medicine injection, participants will be invited for up to four study visits between day 2 and 14 after the injection. This will happen only once during pregnancy, and once during the breastfeeding period to collect a few drops of blood on special filter paper card from the finger using safety lancet. A few drops of breastmilk will also be collected. Immediately after delivery, a few drops of blood will be collected from the mother, umbilical cord and the baby heel.

The investigators will use these samples to determine the amount of the drug in the body during pregnancy and compare this to the amount during the breastfeeding period. Additionally, every month during the third trimester, and during the first 3 months postpartum, participants will complete a questionnaire (using the Liverpool University Neuroleptic Side Effect Scale) to document how they are feeling. Clinical improvement will be documented by the primary care provider using the Clinical Global Impressions Scale.

Findings from this study are expected to help healthcare providers to understand these drugs better so that they can make informed decisions about if and how to use these drugs in women who become pregnant or are breastfeeding.

DETAILED DESCRIPTION:
Primary Objectives

1. To determine the magnitude of changes (if any) in the pharmacokinetics of selected LAIAs during pregnancy and assess the extent of fetal exposure at delivery.
2. To describe breastmilk pharmacokinetics of selected LAIAs and the extent of breastfed infant exposure.

Secondary Objectives

1. To assess safety and clinical outcomes following LAIA use during pregnancy and postpartum.
2. To explore sources of variability in maternal and fetal/breastfed infant LAIA exposure.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant or breastfeeding.
* If pregnant, plans to deliver within the facility.
* Diagnosis of schizophrenia, mania or other psychoses.
* Prescription of long-acting injectable antipsychotic (Risperidone, Paliperidone palmitate, Fluphenazine decanoate, Flupenthixol decanoate and Zuclopenthixol decanoate) as maintenance therapy started before study entry.
* Scheduled to receive at least one injection before delivery (if pregnant) or before week 12 postpartum (if breastfeeding).
* At least 18 of age at study entry.

Exclusion Criteria:

* Unable to understand study information.
* Unable to provide written informed consent.
* Known hypersensitivity to study medication.
* Record of poor medication adherence.
* Personal circumstances will not allow completion of the schedule of study activities.
* Concurrent use of agents with known or uncertain interaction with study drug.
* Currently experiencing severe pregnancy related complications

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant and postpartum women, at least 18 years old receiving maintenance dose of long-acting injectable antipsychotics (LAIA).
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Minimum plasma drug concentration (Cmin) during pregnancy and postpartum | During gestation weeks 33-36 and weeks 9-12 weeks postpartum
  Determined from sampling at the end of a dosing interval during pregnancy, and postpartum
Minimum breastmilk drug concentration (Cmin) | During weeks 9-12 weeks postpartum
  Determined from sampling at the end of a postpartum dosing interval
Maximum plasma drug concentration (Cmin) during pregnancy and postpartum | During gestation weeks 33-36 and weeks 9-12 weeks postpartum
  Highest concentration during a dosing interval during pregnancy, and postpartum
Maximum breastmilk drug concentration (Cmin) | During weeks 9-12 weeks postpartum
  Highest concentration during a postpartum dosing interval
Area under the plasma concentration-time curve (AUC) | During gestation weeks 33-36 and weeks 9-12 weeks postpartum
  For assessment of overall drug exposure in plasma
Area under the breastmilk concentration-time curve (AUC) | During weeks 9-12 weeks postpartum
  For assessment of overall drug exposure in breastmilk
Breastfed infant to maternal plasma LAIA concentration ratio | During weeks 9-12 weeks postpartum
  To determine the level of breastfed infant LAIA exposure and elimination
Newborn to maternal plasma LAIA concentration ratio | As soon as possible after delivery
  To determine the extent of in utero fetal drug exposure and elimination

SECONDARY OUTCOMES:
LAIA associated symptoms | From gestation week 28 to postpartum week 12
  To monitor LAIA side effects during and postpartum using the Liverpool University Neuroleptic Side Effect Rating Scale (LUNSERS)
Clinical improvement | From gestation week 28 to postpartum week 12
  To monitor illness severity, improvement and LAIA efficacy during pregnancy and postpartum using the Clinical Global Impressions Scale.
Single nucleotide polymorphisms in drug disposition genes | From gestation week 28 to postpartum week 12
  To explore genetic sources of interindividual variability in maternal and fetal/breastfed infant drug exposure

CONTACTS AND LOCATIONS:
Overall Officials: Adeniyi Olagunju, PhD, Study Chair — University of Liverpool
Locations (6):
- Nigeria (6):
  - Federal Medical Centre, Makurdi, Benue State
  - Federal Neuropsychiatric Hospital, Kaduna, Kaduna State
  - Federal Neuropsychiatric Hospital, Yaba, Lagos
  - Neuropsychiatric Hospital, Abeokuta, Ogun State
  - Neuropsychiatric Specialist Hospital, Akure, Ondo State
  - Obafemi Awolowo University Teaching Hospital, Ile-Ife, Osun State